CLINICAL TRIAL: NCT02380885
Title: Randomized Controlled Trial of Social Cognition Training and Therapeutic Alliance Focused Therapy for Persons With Severe Mental Illness
Brief Title: RCT Social Cognition Training and Therapeutic Alliance Focused Therapy for Persons With Severe Mental Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bar-Ilan University, Israel (Other)
Collaborators: University of Haifa (Other); Israel Science Foundation (Other)
Responsible Party: Principal Investigator, Ilanit Hasson-Ohayon, Prof. Ilanit Hasson-Ohayon, Bar-Ilan University, Israel
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SCIT3C
Record Dates: First submitted 2015-03-01; First posted 2015-03-05 (Estimated); Results first posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Mental Disorders
Keywords: severe mental illness; social cognition; intervention
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Social Cognition and Interaction Trainin (Experimental): Social Cognition and Interaction Training: psychosocial group intervention
  Interventions: Behavioral: SCIT
- Therapeutic Alliance Focused Therapy (Experimental): Therapeutic Alliance Focused Therapy
  Interventions: Behavioral: TAFT
- Treatment as Usual (No Intervention): Treatment as Usual

INTERVENTIONS:
Behavioral: SCIT — psychosocial group intervention
  Other Names: Social Cognition and Interaction Training
  Arms: Social Cognition and Interaction Trainin
Behavioral: TAFT — psychosocial group intervention
  Other Names: Therapeutic Alliance Focused Therapy
  Arms: Therapeutic Alliance Focused Therapy

SUMMARY:
The study evaluates the effectiveness of the social cognition and interaction training (SCIT), in comparison to both therapeutic alliance focused therapy (TAFT) and treatment as usual (TAU) among persons with severe mental illness. Study purpose: 1) Assess the effectiveness of the SCIT and TAFT interventions, 2) Assess the processes that putatively contribute to the SCIT and TAFT outcomes. Method: A Randomized Controlled Trial (RCT) with approximately one hundred and fifty persons with severe mental illness will be carried out in different psychiatric rehabilitation units and clinics in Israel. To assess the relative effectiveness of the SCIT and TAFT interventions with persons with severe mental illness, both interventions will be compared to treatment as usual (TAU). Clinicians will be trained in both interventions, and outcome measures, including social quality of life and social functioning, as well as mediating processes, including the identification of affective states, ToM, attribution errors and therapeutic alliance, will be assessed. Cognitive functioning and symptom severity will be treated as covariates. Statistical analyses will include analysis of variance which takes into consideration attrition, effect size, mediation processes and covariates.

DETAILED DESCRIPTION:
Social cognition has become an important treatment target for people with schizophrenia since it has been found to be a strong predictor of functional outcome. Social Cognition and Interaction Training (SCIT) is a manualized, group-based intervention that was developed to address the three core deficits in social cognition associated with severe mental illness: emotion perception, Theory of Mind (ToM), and attributional style. SCIT has demonstrated efficacy in improving social cognition and social functioning in both inpatient and outpatient samples. In addition, evidence also shows that the therapeutic alliance is related to various treatment outcomes. Thus, both the SCIT and a therapeutic alliance focused therapy (TAFT) may both affect social cognition and social function, but through different pathways. TAFT was chosen, as comparison to the SCIT, in order to control for interpersonal relationship variables. In this way, the proposed study will evaluate empirically whether the specific techniques for ameliorating the social cognition of persons with severe mental illness that make-up the SCIT enhance social functioning beyond what is achieved through the effective interpersonal ingredients of the therapeutic alliance. Study purpose: 1) Assess the effectiveness of the SCIT and TAFT interventions, 2) Assess the processes that putatively contribute to the SCIT and TAFT outcomes. Method: A Randomized Controlled Trial (RCT) with one hundred and fifty persons with severe mental illness will be carried out in different psychiatric rehabilitation units and clinics in Israel. To assess the relative effectiveness of the SCIT and TAFT interventions with persons with severe mental illness, both interventions will be compared to treatment as usual (TAU). Clinicians will be trained in both interventions, and outcome measures, including social quality of life and social functioning, as well as mediating processes, including the identification of affective states, ToM, attribution errors and therapeutic alliance, will be assessed. Cognitive functioning and symptom severity will be treated as covariates. Statistical analyses will include analysis of variance which takes into consideration attrition, effect size, mediation processes and covariates.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of severe mental disorders (schizophrenia, schizoaffective, bi-polar, depression).
* Ability to provide informed consent.
* Ability to read and write in Hebrew.

Exclusion criteria:

* Co-morbid nuerological condition.
* Hospitalization in the last 6 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ilanit Hasson-Ohayon, Principal Investigator — Department of Psychology, Bar-Ilan University
Locations (5):
- Israel (5):
  - Abarbanel center for mental health, Bat Yam
  - Summit rehabilitation center, Jerusalem
  - Shel Organization, Petah Tikva
  - Enosh, Tel Aviv
  - Keeneret, Tiberias

REFERENCES:
- [Derived] Hasson-Ohayon I, Mashiach-Eizenberg M, Lavi-Rotenberg A, Roe D. Randomized Controlled Trial of Adjunctive Social Cognition and Interaction Training, Adjunctive Therapeutic Alliance Focused Therapy, and Treatment As Usual Among Persons With Serious Mental Illness. Front Psychiatry. 2019 Jun 11;10:364. doi: 10.3389/fpsyt.2019.00364. eCollection 2019. PMID 31244686

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 158 participants participated in the study (158 participants were randomized into three groups).
  Data were collected between the years 2014 and 2018 from four psychiatric rehabilitation agencies.
Groups:
- SCIT: Social Cognition and Interaction Training: psychosocial group intervention
  SCIT: psychosocial group intervention
- TAFT: Therapeutic Alliance Focused Therapy
  TAFT: psychosocial group intervention
- TAU Group: Treatment as Usual
Period: Overall Study
Arm/Group | SCIT | TAFT | TAU Group
Started | 62 | 58 | 38
Completed | 23 | 20 | 20
Not Completed | 39 | 38 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SCIT | TAFT | TAU Group | Total
Number analyzed (Participants) | 23 | 20 | 20 | 63
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 38.9 (11) | 41.4 (12.2) | 39.7 (9.4) | 39.94 (11)
Sex/Gender, Customized [Number; unit: participants]
  male | 12 | 14 | 15 | 41
  female | 11 | 6 | 5 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 23 | 20 | 20 | 63
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Israel | 23 | 20 | 20 | 63
The Face Emotion Identification Task (FEIT) [Mean (Full Range); unit: units on a scale] | 12.83 [0 to 19] | 12.42 [0 to 19] | 11.55 [0 to 19] | 12.29 [0 to 19]

OUTCOME MEASURES:

1. Primary Outcome: The Face Emotion Identification Task (FEIT)
Description: A widely used measure of emotion perception and is indexed by the total number of correctly identified emotions out of nineteen pictured faces (higher number indicates better emotion identification).
Time Frame: This outcome measure was assessed at baseline (Pre-intervention) and at 6 months later (Post-intervention).
Population: Each participant underwent a baseline evaluation prior to his participation of one of the groups (=PRE group), and underwent another evaluation at the end of the group intervention (=POST group, at 6 months)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SCIT | TAFT | TAU Group
Number analyzed (Participants) | 23 | 20 | 20
score on a scale
  PRE group intervention | 12.83 (2.86) | 12.47 (3.71) | 11.55 (3.20)
  POST group intervention | 13.65 (2.71) | 13.65 (3.45) | 12.00 (3.73)

2. Primary Outcome: Faux-Pas Task
Description: The Faux Pas Task is a social cognition assessment tool that measures the ability to detect and understand social faux pas - situations where someone says something they shouldn't have said because they didn't know or realize certain information. Faux-Pas task in its Hebrew version (Shamay-Tsoory, Tomer, Berger, Goldsher, & Aharon-Peretz, 2005) was used to assess TOM. It consist of 10 stories in which a faux pas has occurred and 10 control stories. It assesses emotional and cognitive attributions and the score for each story ranged between 0 to 7. After each story the participants are asked six questions regarding the recognition of faux-pas (understanding the mental state of speaker and listener, understanding the emotional state of the listener). The total score ranges from 0 to 70, when higher scores indicate better ability to detect social mistakes.
Time Frame: This outcome measure was assessed at baseline (Pre-intervention) and at 6 months later (Post-intervention).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SCIT | TAFT | TAU Group
Number analyzed (Participants) | 23 | 20 | 20
score on a scale
  PRE group intervention | 30.79 (8.19) | 30.11 (6.84) | 27.95 (8.11)
  POST group intervention | 34.41 (5.51) | 31.89 (7.98) | 29.20 (8.51)

3. Primary Outcome: Ambiguous Intentions Hostility Questionnaire (AIHQ)
Description: The AIHQ is a measure of attributional style for situations with negative outcomes and ambiguous causality.
  Participants are asked to read each of five vignettes, to imagine that the scenario is happening to her or him, and to write down the reason why the other person acted the way he did toward the participant. Two independent raters subsequently code this written response for the purpose of computing a "hostility bias." The participant then rates the degree to which he or she thinks the other person performed the action on purpose, how angry this action would make the participant feel, and how much the participant would blame the other person.
  Four scales that are calculated: Hostility Bias, Blame Score, Aggression Bias, Intentionality Bias (each is a 5-point Likert scale) .
  In the total scores, each scale can be range from 0 (min) to 25 (max), with higher scores indicating greater attribution of hostile intent, blame, or aggressive response tendencies.
Time Frame: This outcome measure was assessed at baseline (Pre-intervention) and at 6 months later (Post-intervention).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SCIT | TAFT | TAU Group
Number analyzed (Participants) | 23 | 20 | 20
score on a scale
  Hostility bias - pre group intervention | 10.93 (3.50) | 12.63 (4.20) | 11.64 (3.70)
  Hostility bias - post group intervention | 10.19 (2.34) | 11.64 (4.50) | 12.06 (3.61)
  Intentionality score - pre | 12.49 (3.31) | 12.58 (4.66) | 12.42 (3.76)
  Intentionality score - post | 11.69 (2.09) | 11.05 (4.78) | 12.30 (2.96)
  Anger score - pre | 14.9 (4.21) | 14.68 (5.52) | 12.66 (4.50)
  Anger score - post | 13.53 (3.39) | 12.47 (5.64) | 13.47 (5.26)
  Blame score - pre | 14.29 (4.09) | 14.16 (5.92) | 13.05 (4.50)
  Blame score - post | 13 (3.61) | 13 (5.73) | 13.63 (4.42)

4. Primary Outcome: Social Skill Performance Assessment
Description: The SSPA is a verbal role-play assessment in which the subject participates in two 3-minute role-play conversations ("scenes") with the assessor on pre-determined topics (e.g. "Your landlord has not fixed a leak that you told him about last week, and now you are calling him on the phone to follow-up."). Role-plays are tape-recorded and rated by independent coders. Each one of the 17 domains is rated on a 5-point Likert-type scale. Thus, the total score for the task can be ranged from 0 (min) to 85 (max), with higher scores signifying greater social skills.
  The SSPA has good face validity as a social skill measure and among individuals with schizophrenia it shown excellent inter-rater reliability, good test-retest reliability, and good convergent validity with a measure of activities of daily living. It is a 5-point Likert-type scale with higher scores signifying greater social skill.
Time Frame: This outcome measure was assessed at baseline (Pre-intervention) and at 6 months later (Post-intervention).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SCIT | TAFT | TAU Group
Number analyzed (Participants) | 23 | 20 | 20
score on a scale
  PRE group intervention | 47.13 (13.3) | 48.90 (13.4) | 54 (16)
  POST group intervention | 52.39 (16.6) | 50.20 (12.7) | 49.70 (16.2)

5. Secondary Outcome: Wisconsin Social Quality of Life Scale.
Description: The Wisconsin Quality of Life Scale (W-QLI) is a multidimensional assessment tool designed to measure quality of life, particularly for individuals with mental illness.
  The scores range from 0 to 7, with the higher score indicating higher social QoL.
Time Frame: This outcome measure was assessed at baseline (Pre-intervention) and at 6 months later (Post-intervention).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SCIT | TAFT | TAU Group
Number analyzed (Participants) | 23 | 20 | 20
score on a scale
  PRE group intervention | 4.48 (1.22) | 5.22 (1.35) | 4.78 (1.40)
  POST group intervention | 4.61 (1.31) | 5.23 (1.53) | 4.77 (1.32)

ADVERSE EVENTS:
Time Frame: 2 years.
Description: the definition of adverse event and/or serious adverse event does not differ from the clinicaltrials.gov Definitions.
Groups:
- TAU - Treatment as Usual: Treatment as Usual
Arm/Group | SCIT | TAFT | TAU - Treatment as Usual
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/23 | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-10): https://cdn.clinicaltrials.gov/large-docs/85/NCT02380885/Prot_SAP_001.pdf